CLINICAL TRIAL: NCT05280249
Title: The Effects of Green Exercise Program Consisting of 12-week Aerobic and Resistance Exercises on Sleep Quality, Alexithymia, Anxiety and Depression in Elderly People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07.03.2022
Record Dates: First submitted 2022-03-07; First posted 2022-03-15 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-03

CONDITIONS: Elderly; Exercise
Keywords: elderly; exercise; Affective Symptoms; anxiety; depression
MeSH Terms: conditions — Motor Activity; Affective Symptoms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Parallel Assignment Randomized
Who Masked: Outcomes Assessor
Masking Description: Evaluations will be made by an impartial researcher who was not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Both aerobic and resistance exercises in the green exercise concept (Experimental): Green exercise is a type of exercise done outdoors. It is an advantageous type of exercise in benefiting from sunlight and reducing anxiety. Participants in this group will be given aerobic and resistance exercises in the open air. For 20 participants who met the inclusion criteria, first 10 minutes of warm-up exercises, then 20 minutes of moderate-intensity (65% of heart rate) walking, followed by 15 minutes of low-intensity (50% of the maximum repetitions) resistance exercises will be trained in the presence of a physiotherapist. resistance exercises will be performed for shoulder flexors and abductors, elbow flexors and extensors, hip flexors and extensors, knee flexors and extensors, hip abductor muscle groups. At the end of each session, 5 minutes of stretching exercises will also be trained.
  Interventions: Other: both aerobic and resistance exercises in the green exercise concept
- Control group (No Intervention): The exercise program will not be implemented. Evaluations will be made at the beginning and end of the study.

INTERVENTIONS:
Other: both aerobic and resistance exercises in the green exercise concept — Green exercise is a type of exercise done outdoors. It is an advantageous type of exercise in benefiting from sunlight and reducing anxiety. Participants in this group will be given aerobic and resistance exercises in the open air.
  Arms: Both aerobic and resistance exercises in the green exercise concept

SUMMARY:
The aim of this study is to investigate the effects of combination of aerobic and resistance exercises in the green exercise concept on depression, anxiety, alexithymia and sleep quality of elderly individuals. Elderly individuals over the age of 65 will be included in the study. Two groups of 20 people each will take part in the study. One group will be given aerobic and resistance exercises for 12 weeks, 2 days a week in the green exercise concept, the other group will be the control group and will not be included in the exercise program. Participants will be evaluated twice, at the beginning of the study and at the end of 12 weeks.

DETAILED DESCRIPTION:
Forty volunteer participants aged 65 years over will be included in the study. Participants will be randomly divided into two groups as experimental and control group. While experimental group will receive both aerobic and resistance exercises and control group will receive no exercise. Exercises will be held in an open and green area. Depression, anxiety, alexithymia and sleep quality of elderly individuals will be evaulated at the beginning of the treatment and at the end of the twelfth week. The exercise program will be done for 12 weeks, 2 days a week.

ELIGIBILITY:
Inclusion Criteria:

* people aged over 65 years
* Be fit to participate in exercise program after the first cardiac examination by the physician
* Having a score above 24 in the Minimental Test

Exclusion Criteria:

* Having neuromuscular disease
* Serious medical condition (for example, advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.)
* Having an orthopedic disease that interferes with walking
* Having a score below 24 in the Minimental Test

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-09-12 (Estimated); Study Completion 2022-10-17 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Change from baseline sleep quality at week 12.
  Sleep quality will be evaulated with Pittsburg Sleep Quality Index (PUKI). PUKI was developed by Buysee et al. in 1989 and provides a quantitative measure of sleep quality. It contains a total of 24 questions. Each item is scored between 0-3 points. It has 7 components (subjective sleep quality, sleep duration, sleep disturbance, sleep latency, habitual sleep efficiency, sleep medication use, daytime dysfunction). The sum of the scores of these seven components gives the total index score. High scores indicate poor sleep quality.
Anxiety | Change from baseline anxiety level at week 12.
  Anxiety will be evaluated with Geriatric Anxiety Scale. It is a self-filled scale developed for the elderly, observing anxiety symptoms, having somatic, cognitive and affective subscales. It is a 4-point Likert scale scored between 0-3 and consists of 30 questions in total. Items between 24 and 28 are not included in the total score, clinicians use these items to determine the domain of anxiety. The total score ranges from 0 to 75. A high score indicates a high level of anxiety.
Depression | Change from baseline depression level at week 12.
  Depression will be assessed with the Geriatric Depression Scale. GDS is a self-reported scale consisting of 30 questions and asked to be answered in a yes/no format. In scoring the scale, 1 point is given for each answer in favor of depression, 0 point is given for the other answer, and the total score is accepted as the depression score. The scores that can be obtained from the scale are between 0-30.
Alexithymia | Change from baseline alexithymia level at week 12.
  Alexithymia, also called emotional deafness, is a psychopathology characterized by difficulties in understanding, defining and expressing their own emotions. Alexithymia will be evaulated Toronto Alexithymia Scale-20. It is a Likert-type scale scored between 1 and 5, and includes 20 questions in total. Items 4,5,10,18 and 19 are reverse scored. Those with a total score of 61 and above are considered to have alexithymia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No